CLINICAL TRIAL: NCT02113410
Title: Effect of Sit 'N' Fit Chair Yoga on Community-Dwelling Elders With Osteoarthritis
Brief Title: Effect of Chair Yoga on Elders With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 420926; 1R15AT007352-01A1 (NIH)
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis (OA)
Keywords: osteoarthritis; Older adults; Sit 'N' Chair Yoga; Pain; Physical Function; Balance; Fatigue; Depression; Life Satisfaction
MeSH Terms: conditions — Osteoarthritis; Pain; Fatigue; Depression; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sit 'N' Fit Chair Yoga (SNFCY) (Experimental): Willing and eligible subjects randomized to Sit 'N' Fit Chair Yoga attended twice-weekly 45-minute yoga sessions for 8 weeks, for a total of 16 sessions.
  Interventions: Behavioral: Sit 'N' Fit Chair Yoga (SNFCY)
- Health Education Program (HEP) (Active Comparator): Willing and eligible subjects randomized to the Health Education Program (HEP) will attended twice-weekly 45-minute health education sessions for 8 weeks, for a total of 16 sessions.
  Interventions: Behavioral: Health Education Program (HEP)

INTERVENTIONS:
Behavioral: Sit 'N' Fit Chair Yoga (SNFCY) — Experimental: Sit 'N' Fit Chair Yoga - a twice-weekly, 8-week yoga program of 45-minute sessions. Active Comparator: Health Education Program (HEP), a twice-weekly, 8-week program of 45-minute sessions
  Arms: Sit 'N' Fit Chair Yoga (SNFCY)
Behavioral: Health Education Program (HEP) — Willing and eligible subjects randomized to the Health Education Program (HEP) attended twice-weekly 45-minute health education sessions for 8 weeks, for a total of 16 sessions.
  Arms: Health Education Program (HEP)

SUMMARY:
The current study is a two-arm randomized controlled clinical trial to test the feasibility of recruiting, randomizing, and having older adults with osteoarthritis (OA) adhere to and safely complete the 8-week Sit 'N' Fit Chair Yoga program and the HEP program (primary objective). Secondary objectives of the study were to determine the effect of the Sit 'N' Fit Chair Yoga Program to reduce levels of pain; improve physical function, psychosocial function, and life satisfaction in adults over 65 years of age who were unable to participate in standing exercise. Participants at two sites were randomly assigned to either the intervention group (Sit 'N' Fit Chair Yoga) or attention control group (Health Education Program). Data collectors were blinded to group assignments. Data were collected prior to the intervention (baseline), after 4 weeks, and after 8 weeks. Follow-up data were collected after 1 month and after 3 months after completion of the intervention to measure the extent to which effects of the intervention continue. Evaluations were include physical measures and self-report measures.

DETAILED DESCRIPTION:
Consenting Procedure

An informed consent was obtained from the participants, followed by screening for eligibility. The Project Directors, the PIs, or data collectors discussed the project and obtained the informed consent. At the two study sites, all participants lived independently and were able to sign informed consent. If changes to the study design or program were made, new consents were obtained from all participants after IRB and NCCIH's approval. One copy of the consent was provided to the participant and one copy was kept in a file in the PIs' office in a locked file cabinet. An ID number was assigned to each participant and placed on the second copy of the consent form.

Randomization: Each participant who met the eligibility criteria and who signed informed consent was given an ID number from that list. An overall list of participants with ID numbers were created by the Project Director as participants are enrolled. Participants were enrolled within the 1-week time frame described in the protocol, the outside statistician sent a randomization pattern to the Project Director at each site. The Project Directors matched the randomization pattern with the list of participants to determine to which arm of the study each participant was assigned.

The study statistician, the two Principal Investigators(PIs), and the two Project Directors were responsible for data management. Dr. Newman and the two PIs reviewed all data collection forms on an ongoing basis for data completeness and accuracy, as well as for protocol compliance. They supervised the Project Directors at each site. All the research members including PIs, Project Directors, data collectors, and yoga and HEP instructors completed safety training. All completed forms, including demographic information, were secured in a locked cabinet in primary statistician office at FAU.

The statistician and his research assistant entered data independently (double data entry) using password-protected access to the SPSS data entry system after data collection period (baseline, 4 weeks, 8 weeks, and 1 month and 3 months after intervention). They compared the databases for data entry error and will check the error rate. All data were backed up on FAU secure servers. The primary statistician (Dr. Newman) cleaned the data and randomly selected 10% of all cases in each data entry batch to check for data entry error. An examination of each statistical model was conducted to examine the normality of the residuals and to look for outliers and overly-influential data points. The PIs met with the primary statistician, the Project Directors, and the RAs on a regular basis to discuss progress in data entry, data analysis and interpretations of the results, and other issues related to data management.

SAFETY ASSESSMENTS:

Study progress and safety were reviewed quarterly. The study statistician, PIs, Project Directors, and Data and Safety Monitoring Committee (DSMC) reviewed AE rates. Progress reports, including participant recruitment, adherence and retention/attrition, were provided to the DSMC following each quarterly review. The quarterly report included a list and summary of adverse events (AE), using ID numbers only. The report was sent to the DSMC of independent monitors and forwarded to the IRB and NCCIH. The IRB reviewed progress of the study annually and the PI sent the final/closing report to IRB in November 2016.

An adverse finding from attending the Chair Yoga session could include increased pain, muscle ache/cramping, fatigue, or any combination of these.

A serious adverse event (SAE) is any AE that results in one or more of the following outcomes regardless of relationship to study intervention:

* A life-threatening event
* Inpatient hospitalization or prolongation of existing hospitalization
* A persistent or significant disability/incapacity
* An important medical event, based on appropriate medical judgment

Measurement Tools:

Ten measurement tools will be used to determine the effect of the Sit N Fit Chair Yoga program and the Health Education Program on the study outcome measures. These tools are:

Western Ontario and McMaster Universities Arthritis Index (WOMAC) PROMIS Pain Interference Scale Gait Speed Six-Minute Walk Test (6MWT) Berg Balance Scale PROMIS Physical Function Short Form PROMIS Fatigue Scale Short Form Life Satisfaction Index for Third Age, Short Form (LSITA-SF) PROMIS Ability to Participate in Social Roles and Activities Short Form PROMIS Emotional Distress-Depression Short Form

Data Analyses

Analyses were performed using SPSS software, version 23.0 (IBM) and HLM 7.01 (SSI International). The Missing Value Analysis function in SPSS was employed to ascertain the extent, randomness, and pattern of missing data. Hierarchical linear models (HLM) were used to analyze change over time for each participant. Depending on the nature of the change function, parameter estimates were calculated for intercept, slope and, if necessary, curvature to create the best predictive model fit. Because HLM shows longitudinal changes as a function of time, the time variable was centered at the baseline. The results for the fixed-effects model were used to report the treatment effects for both 8-week ITT assessment and 3-month post-intervention. The random effects model assessed overall changes in all outcomes over the same time periods.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 years or older
2. living independently in the community and noninstitutionalized at the time of the study
3. self-reported joint pain verified by Dr. McCaffrey and a Project Director (nurse practitioner) to be caused by OA and present in one or more lower extremity joints (hip, knee, foot, or ankle)
4. ability to ambulate independently with or without assistive devices
5. chronic pain at least 15 days of the month for 3 months or longer at a level of at least 4 (moderate pain) on a 0-10 pain bothersomeness scale (0 = no pain to 10 = excruciating pain)
6. self-reported inability to participate in regular yoga or standing exercise due to physical disability, fatigue, fear of falling, or balance problems
7. not currently participating in yoga or any other exercise program
8. ability to understand English or Spanish
9. ability to come to designated site at the scheduled times
10. willingness to be audiotaped during the intervention sessions

Exclusion Criteria:

1. Knee surgery (or knee-arthroscopy) or hip(s) within 12 weeks prior to enrollment, causing pain or functional problems
2. Systemic or intra-articular corticosteroid use within 60 days of the screening visit
3. Serious comorbidity that makes it impossible to participate in the yoga intervention (e.g., heart failure-New York Heart Association (NYHA IV)
4. Require assistance by another person (e.g., holding the arm or walking behind) in order to ambulate 30 feet
5. Participation in yoga or exercise program currently or in the previous 3 months, or planning to participate in yoga or other exercise program during the chair yoga intervention (including 3-month follow-up)
6. Intra-articular steroid injections within 4 weeks of screening
7. Inability to understand or speak English or Spanish
8. Inability to correctly answer questions, complete the demographic data form, and continue with yoga practice for 1 month post intervention. This is measured by asking participants the following questions (Alzheimer's Association's "questions to determine early cognitive impairment) (http://www.alz.org/alzheimers_disease_10_signs_of_alzheimers.asp) as accessed August 27, 2013, as approved by our geriatric content expert, Dr. Joseph Ouslander).

Those who answer three or more of these questions incorrectly are excluded from the study.

1. What is today's date? 2. What day of the week is today? 3. On what street do you live? 4. In what town do you live? 5. In what state is your town? 6. Who is the President? 7. What season of the year is this? 8. What month are we in now? 9. How did you get here today?

Screening Evaluation

All participants must have OA. As diagnostic criteria for OA, the participant must exhibit at least three of the following upon history or physical examination to be considered to have a diagnosis of OA and thus to be eligible to participate in the study:

* Pain in the affected joint
* Morning stiffness that is relieved as the day progresses
* Crepitus on active motion
* Bony tenderness
* Bony enlargement
* Decreased range of motion of joint
* Joint instability upon standing or bending
* Increased pain and fatigue with walking or standing
* The participant must ambulate at least 30 feet without assistance from another person (may use cane, walker, or wheelchair). Those who require personal assistance to ambu-late 30 feet (such as needing to hold an arm or to have someone walk behind for safety) are excluded because they would not be able to complete the 6-Minute Walk or Gait Speed Test.

During the screening of potential participants each person is asked whether he or she is able to participate in standing exercise programs or regular yoga programs. The following questions are asked and people are eligible if they identify any two of the following:

Please check any of the following that you feel unable to do because of balance, pain, fear of falling, fatigue or strength

* Standing for 30-45 minutes
* Bending over toward your toes
* Bending side to side
* Squatting
* Standing on one foot
* Standing, holding your arms outstretched above your head
* Twisting your body side to side

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juyoung Park, Ph. D, Principal Investigator — Florida Atlantic University; Patricia Liehr, Ph.D., Principal Investigator — Florida Atlantic University
Locations (2):
- United States (2):
  - North East Focal Point Senior Center, Deerfield Beach, Florida
  - Douglas Gardens North (Public Housing Facility), Pembroke Pines, Florida

REFERENCES:
- [Derived] Park J, McCaffrey R, Newman D, Liehr P, Ouslander JG. A Pilot Randomized Controlled Trial of the Effects of Chair Yoga on Pain and Physical Function Among Community-Dwelling Older Adults With Lower Extremity Osteoarthritis. J Am Geriatr Soc. 2017 Mar;65(3):592-597. doi: 10.1111/jgs.14717. Epub 2016 Dec 23. PMID 28008603
- [Derived] McCaffrey R, Park J, Newman D. Chair Yoga: Feasibility and Sustainability Study With Older Community-Dwelling Adults With Osteoarthritis. Holist Nurs Pract. 2017 May/Jun;31(3):148-157. doi: 10.1097/HNP.0000000000000184. PMID 27782922

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two settings-a senior housing facility and a senior day center-through an information session conducted at each site by the principal investigators and Project Directors. There were 3 cohorts (waves) in the study. In each cohort, recruitment was started 2 weeks prior to the each intervention.
Groups:
- Health Education Program (HEP): To control for attention and time, HEP participants attended twice-weekly 45-minute sessions for 8 weeks led by health care providers trained by the principal investigators. The instructors received two 4-hour days being trained on HEP teaching instructions and serving as an arbitrator of any disagreements between participants on a certain topic. HEP participants discussed general health education information and specific facts regarding OA; they did not participate in any form of yoga.
- Sit 'N' Fit Chair Yoga: The chair yoga intervention consisted of twice-weekly 45-minute sessions incorporating four components-physical postures, breathing, deep relaxation, and meditation-while using the support of a chair. The yoga instructor at each site was certified by the Yoga Alliance and spent two 8-hour days being trained on the Sit "N" Fit Chair Yoga program by the program developer.
Period: Overall Study
Arm/Group | Health Education Program (HEP) | Sit 'N' Fit Chair Yoga
Started | 65 | 66
Completed | 49 | 63
Not Completed | 16 | 3

BASELINE CHARACTERISTICS:
Groups:
- Sit N Fit Chair Yoga: The chair yoga intervention consisted of twice-weekly 45-minute sessions incorporating four components-physical postures, breathing, deep relaxation, and meditation-while using the support of a chair. The yoga instructor at each site was certified by the Yoga Alliance and spent two 8-hour days being trained on the Sit "N" Fit Chair Yoga program by the program developer.
- Health Education Program: To control for attention and time, HEP participants attended twice-weekly 45-minute sessions for 8 weeks led by health care providers trained by the principal investigators. The instructors received two 4-hour days being trained on HEP teaching instructions and serving as an arbitrator of any disagreements between participants on a certain topic. HEP participants discussed general health education information and specific facts regarding OA; they did not participate in any form of yoga.
- Total: Total of all reporting groups
Arm/Group | Sit N Fit Chair Yoga | Health Education Program | Total
Number analyzed (Participants) | 63 | 49 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 63 | 49 | 112
Age, Continuous [Mean (Standard Deviation); unit: year] | 75.9 (8.2) | 74.5 (6.5) | 75.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 19 | 8 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 26 | 52
  Not Hispanic or Latino | 37 | 23 | 60
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 49 | 112

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Pain Interference
Description: The 8-item PROMIS Pain Inference-Short Form- V. 1.0-8a was administered to measure self-reported consequences of pain on various aspects of the participant's life.Scores can range from 8 (minimum) to 40 (maximum) and higher scores indicate more interference with daily activities. This tool is normed on the U.S. general population, with an average score of 50 and a standard deviation of 10, to report interference within the previous 7 days on 5-point response scale ranging from not at all to very much. This self-report measure was developed by the NIH. NIH has rigorously tested the construct validity and reliability of all of the PROMIS tools and all have been shown to be internally consistent, reliable (reliability = .96 to .99, for PROMIS-PI SF) and valid (construct validity). A higher score represent a severe pain level.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sit 'N' Fit Chair Yoga (SNFCY): Of the 66 participants who were assigned to SNFCY, 2 dropped after randomization but prior to intervention. Thus, 64 started the intervention; however, 1 dropped during the intervention. Sixty three participants completed the intervention. Of 63 participants, 61 completed at least 12 of 16 sessions and provided data at all five data collection points, for a retention rate of 96% (61/63).
- Health Education Program (HEP): Of the 65 participants who were assigned to HEP, 11 dropped after randomization but prior to intervention. Thus, 54 started the intervention; however, 5 dropped during the intervention due to schedule conflict, personal issues, or family illness. Forty nine participants completed the intervention. Of 49 participants, 45 completed at least 12 of 16 sessions and provided data at all five data collection points, for a retention rate of 92% (45/49).
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline | 19.0 (7.3) | 19.1 (8.7)
  4 weeks of the intervention | 18.0 (8.2) | 17.5 (8.3)
  8 weeks of the intervention | 15.1 (7.3) | 18.3 (8.9)
  1 month follow-up | 15.7 (7.6) | 19.1 (8.2)
  3 month follow-up | 15.5 (7.4) | 17.3 (8.9)

2. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The Western Ontario and McMaster Universities Osteoarthritis Index was administered to measure self-reported. The tool, recommended for osteoarthritis clinical trials, is a self-administered scale with 24 questions using a Likert-type scale. The Western Ontario and McMaster Universities Osteoarthritis Index was administered to measure self-reported OA symptoms (pain, stiffness, functional ability). The tool is a self-administered scale with 24 items (pain [5 items], stiffness [2 items], physical function [17 items]). A score range for each subscale for each scale (minimum-maximum) is Pain 0-20, stiffness 0-8, physical function 0-68. Higher scores indicate worse pain, stiffness, and functional limitations. For this study, we used a subscale of pain (5 items), stiffness (2 items), physical function (17 items). A total score of all subscales can range from 0 (minimum) to 96 (maximum). The WOMAC demonstrated a Cronbach's alpha of .95 for persons with OA.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline | 6.6 (3.7) | 7.2 (4.4)
  4 weeks | 5.7 (3.5) | 5.8 (4.0)
  8 weeks (post intervention) | 4.5 (3.3) | 6.4 (4.6)
  1-month follow up | 4.6 (3.5) | 5.7 (4.4)
  3-month follow up | 4.6 (3.6) | 5.5 (4.4)

3. Secondary Outcome: PROMIS Physical Function
Description: The PROMIS Physical Function Short Form-V 1.0-12a was administered to measure physical function. The domain of physical function assesses self-reported ability rather than actual performance of physical activities. Scores can range from 7 (minimum) to 60 (maximum). The higher scores represent better physical function.This includes functioning of upper extremities (dexterity), lower extremities (mobility), and central regions (neck back), as well as instrumental activities of daily living. Each question has five response options, ranging in value from 1 (unable to do) to 5 (able to do without any difficulty).
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline | 37.0 (7.5) | 35.2 (8.4)
  4 weeks of the intervention | 37.4 (6.5) | 36.6 (9.4)
  8 weeks of the intervention | 38.2 (7.1) | 36.0 (9.2)
  1 month follow-up | 38.5 (6.5) | 38.0 (8.3)
  3 month follow-up | 39.4 (7.3) | 37.0 (8.4)

4. Secondary Outcome: Gait Speed Test
Description: The Gait Speed Test was used to measure physical function. Gait speed measurement is considered highly reliable in older adults without known impairments that should affect gait. For measuring gait speed, the unit of measurement is the second. Intrarater reliability (N = 19-24) and test-retest reliability (N = 19-41) have been reported as high (ICC = .90-.96, r = 89-100). The Pearson correlation coefficient is r = .93 and ICC = .78 for test-retest reliability for gait speed in older adults.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: time (second)
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
time (second)
  Baseline | 8.6 (4.0) | 7.8 (3.0)
  4 weeks of the intervention | 8.2 (3.3) | 9.0 (4.6)
  8 weeks (post intervention) | 8.1 (2.9) | 8.3 (3.4)
  1 month follow-up | 7.7 (2.3) | 8.0 (3.1)
  3 month follow-up | 7.7 (3.1) | 7.7 (3.4)

5. Secondary Outcome: Berg Balance Scale
Description: The Berg Balance Scale was administered to measure changes in balance function. The performance-based Berg Balance Scale contains 14 items applying a 5-point scale for each item (0 = lowest level of function to 4 = highest level of function); scores range from 0 to 56. Higher scores indicate higher fall risk. The Berg Balance Scale is the gold standard assessment of balance, obtaining good to excellent intra-rater reliability (ICC = 0.68-0.99) and interrater reliability (ICC = 0.88-0.98) and good internal validity.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
scores on a scale
  baseline | 31.4 (7.9) | 30.6 (8.6)
  4 weeks of the intervention | 34.7 (7.3) | 31.5 (10.3)
  8 weeks (post intervention) | 35.0 (6.4) | 33.1 (7.6)
  1 month follow-up | 35.1 (7.9) | 33.2 (9.3)
  3 month follow-up | 35.0 (8.4) | 32.5 (8.7)

6. Secondary Outcome: 6-Minute Walk Test
Description: The 6-Minute Walk Test was administered to measure changes in exercise tolerance in participants. The tool measured the distance(yards) a participant walked in 6 minutes on a hard and flat surface. Less distances (yards) covered in 6 minutes indicate lower function.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: yards
Groups:
- Sit 'N' Fit Chair Yoga (SNFCY): Of the 66 participants who were assigned to SNFCY, 2 dropped after randomization but prior to intervention. Thus, 64 started the intervention; however, 1 dropped during the intervention. Sixty three participants completed the intervention. Of 63 participants, 61 completed at least 12 of 16 sessions (Figure 1) and provided data at all five data collection points, for a retention rate of 96% (61/63).
- Health Education Program (HEP): Of the 65 participants who were assigned to HEP, 11 dropped after randomization but prior to intervention. Thus, 54 started the intervention; however, 5 dropped during the intervention due to schedule conflict, personal issues, or family illness. Forty nine participants completed the intervention. Of 49 participants, 45 completed at least 12 of 16 sessions (Figure 1) and provided data at all five data collection points, for a retention rate of 92% (45/49).
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
yards
  baseline | 205.6 (142.6) | 204.5 (155.5)
  4 weeks of the intervention | 223.2 (154.7) | 189.4 (132.2)
  8 weeks (post intervention) | 218.5 (168.0) | 205.0 (139.6)
  1 month follow-up | 213.4 (144.7) | 224.7 (133.7)
  3 month follow-up | 207.0 (149.6) | 219.6 (132.8)

7. Secondary Outcome: PROMIS Emotional Distress-Depression (Short Form)
Description: The PROMIS Emotional Distress and Depression-V 1.0-Short Form-8a was administered o measure depressive symptoms. The tool has a 5-point scale for each item (1 = Never to 5 = Always); scores can range from 8 to 40. Higher scores indicate higher levels of depression and emotional distress.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
scores on a scale
  baseline | 14.3 (5.7) | 14.2 (6.0)
  4 weeks | 13.5 (5.4) | 12.8 (5.6)
  8 weeks (post intervention) | 12.5 (5.3) | 13.0 (6.4)
  1 month follow-up | 14.1 (6.2) | 12.9 (5.9)
  3 month follow-up | 12.6 (5.1) | 13.2 (6.4)

8. Secondary Outcome: PROMIS Fatigue Scale
Description: The PROMIS Fatigue scale was administered to evaluate a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that decreases ability to execute daily activities and to function normally in family or social roles.It ranges 8-40 and higher scores indicate higher level of fatigue.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: score on the scale
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
score on the scale
  baseline | 20.1 (7.4) | 20.5 (8.3)
  4 weeks of the intervention | 19.6 (6.6) | 20.4 (8.0)
  8 weeks (post intervention) | 17.8 (7.1) | 20.4 (7.9)
  1 month follow-up | 18.1 (6.5) | 19.2 (7.4)
  3 month follow-up | 17.9 (6.9) | 19.3 (8.3)

9. Secondary Outcome: PROMIS Ability to Participate in Social Activities
Description: The PROMIS Ability to Participate in Social Activities-V 2.0- SF-8a was administered to measure the perceived ability to perform usual social roles and activities. Items are worded negatively in terms of perceived limitations (5 = Never to 1 = Always), but responses are reverse-coded .Scores can range from 8 to 40; higher scores indicate lower ability to participate in social roles.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: score on the scale
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
score on the scale
  baseline | 27.2 (8.1) | 27.8 (10.0)
  4 weeks of the intervention | 28.5 (7.8) | 26.5 (9.7)
  8 weeks (post intervention) | 29.9 (7.8) | 27.2 (9.5)
  1 month follow-up | 28.5 (7.7) | 28.0 (8.4)
  3 month follow-up | 29.8 (7.4) | 28.6 (9.1)

10. Secondary Outcome: Life Satisfaction Index-Short Form (LSITA-SF)
Description: The Life Satisfaction Index-Short Form was administered to measure general life satisfaction in participants. The 12-item index offers a 6-point scale for each item (1 = strongly agree to 6 = strongly disagree; for Items 2, 4, 5, and 6, the responses are reversed. It ranges 12 (minimum)-72 (maximum); higher scores indicate higher level of life satisfaction. Reliability of this instrument when used with 654 older adults produced a Cronbach's alpha of .95, with a goodness of fit of > .90. It has a correlated reliability of .90 with the long form.
Time Frame: 6 months
Population: Community-dwelling Older adults (age 65 years or older) who are diagnosed with osteoarthritis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline | 38.9 (9.1) | 38.4 (9.3)
  4 weeks of the intervention | 38.4 (8.6) | 36.8 (9.3)
  8 weeks (post intervention) | 38.1 (9.6) | 36.5 (8.8)
  1 month follow-up | 39.8 (9.2) | 36.5 (9.1)
  3 month follow-up | 37.7 (9.3) | 37.2 (9.6)

ADVERSE EVENTS:
Time Frame: 6 months for each wave
Description: 131
Groups:
- Sit 'N' Fit Chair Yoga (SNFCY): There were no adverse events or serious adverse events associate with SNFCY.
- Health Education Program (HEP): There were no adverse events or serious adverse events associate with HEP.
Arm/Group | Sit 'N' Fit Chair Yoga (SNFCY) | Health Education Program (HEP)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/49
Other Adverse Events (participants affected / at risk) | 0/63 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No